CLINICAL TRIAL: NCT05518695
Title: A Randomized, Double-Blind, Phase I Clinical Study to Evaluate the Pharmacokinetics of BAT2022 in Healthy Chinese Subjects
Brief Title: Evaluate the Pharmacokinetics of BAT2022 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-2022-001-CR
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — BAT2022; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1/100mg (Experimental): Drug:BAT2022 for Intravenous fluids 100mg
  Interventions: Drug: BAT2022
- A2/300mg (Experimental): Drug:BAT2022 for Intravenous fluids 300mg
  Interventions: Drug: BAT2022
- A3/1000mg (Experimental): Drug:BAT2022 for Intravenous fluids 1000mg
  Interventions: Drug: BAT2022
- A4/1500mg (Experimental): Drug:BAT2022 for Intravenous fluids 1500mg
  Interventions: Drug: BAT2022

INTERVENTIONS:
Drug: BAT2022 — Eight healthy subjects are planned to be enrolled in each group, 6 on the investigational product and 2 on placebo. Subjects will be randomized (3:1) to receive a single intravenous injection of BAT2022 for Injection or 5% glucose injection. Sentinel dosing will be performed for subjects in each group.Two subjects in each group who have received the first dose will be randomized (1:1) to either the test group or placebo group. After observation for 24 h and the drug is safe and well tolerated, the remaining subjects in this group will be randomized (5:1) to either the test group or placebo group.
  Other Names: BAT2022 for Injection (bispecific neutralizing antibody targeting the receptor binding domain (RBD) of spike of SARS-CoV-2)

SUMMARY:
To evaluate the safety and tolerability of BAT2022 in healthy subjects.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled, dose-escalation clinical study to evaluate the pharmacokinetics, safety, tolerability, immunogenicity and pharmacodynamics of BAT2022 for Injection in healthy subjects.

ELIGIBILITY:
: Inclusion Criteria:

1. Subjects who have signed the informed consent form prior to the study and have a full understanding of the content, process and possible adverse reactions;
2. Subjects who are willing and able to follow the visit and treatment specified in this study;
3. Subject (including partner) who is willing to have no pregnancy plan or sperm donation plan within the following 6 months (i.e., within 6 months after administration of the investigational product) and voluntarily take effective contraceptive measures;
4. Healthy male or female subjects aged 18 ~ 55 years (inclusive);
5. Subjects with body weight of 50 kg ~ 100 kg (inclusive);
6. Subjects with normal or abnormal physical examination without clinical significance;

Exclusion Criteria:

1. Subjects who have smoked more than 5 cigarettes per day three months prior to Screening;
2. Any subject with a current or past serious allergic reaction to food or drug, or serious allergic or allergic reaction to human, humanized or mouse monoclonal antibody;
3. Subjects with a history of alcoholism (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of liquor, or 125 mL of wine);
4. Subjects who have donated blood or had massive blood loss (>450 mL) within three months prior to screening, or intend to donate blood or undergo surgery during the study;
5. Subjects who have taken any prescription drug, over-the-counter drug, any vitamin products or herbal medicines 28 days prior to Screening;
6. Subjects who have significant changes in diet or exercise habits 2 weeks prior to screening or from screening to administration;
7. Subjects who have used any biological products within 3 months prior to screening;
8. Subjects with clinical significance of abnormal heart assessed using Color Doppler echocardiography
9. Subjects with clinical significance of abnormal laboratory findings (hematology, urinalysis, serum chemistry, coagulation function, virology of infectious diseases and pregnancy test for women of childbearing age), or other clinical findings suggestive of the following disorders with clinical relevance (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immune, psychiatric or cardiovascular and cerebrovascular diseases);
10. Subjects with clinical significance of abnormal (as judged by the investigator) ECG, or QTcF > 450 ms (allowed to be repeated for once);
11. Subjects with acute illness or concomitant medication from screening to prior to administration of the investigational product;
12. Subjects with positive urine drug screen, or subjects with a history of drug abuse or drug use in the past 5 years;
13. Subjects who have taken any alcohol-containing products within 48 hours prior to administration of the investigational product, or who are unable to limit alcohol consumption as required during the course of the study;
14. Subjects with current or previous malignant tumours;
15. Subjects with a history of hypertension or systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg at screening/baseline;
16. Subjects with liver disorder who are judged by the investigator as inappropriate for enrollment;
17. Subjects with abnormal focal shadows on chest radiograph, including but not limited to active pulmonary tuberculosis;
18. Subjects who have participated in drug clinical study within three months prior to the first dose of the investigational product, or planned to participate in other drug clinical study during the study;
19. Subjects who are considered by the investigator as inappropriate for enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | DLT observation period is 7 days postdose.
  Grade ≥3 AEs in this criteria are defined as dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) | DLT observation period is 7 days postdose.
  it is determined that ≥ 50% of subjects have experienced a DLT as defined in this protocol

CONTACTS AND LOCATIONS:
Overall Officials: Weiyong Li, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital Tong Ji Medical College University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No